CLINICAL TRIAL: NCT06707675
Title: Chronotype and Quality of Life in Patients with Myofascial Pain Syndrome, a Cross-Sectional Study
Brief Title: Chronotype and Myofascial Pain Syndrome,
Status: Not yet recruiting | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, Ass. Prof., Afyonkarahisar Health Sciences University
Other Study IDs: SAMAS
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Myofascial Pain Syndrome, Diffuse
MeSH Terms: conditions — Fibromyalgia | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MPS: Patients aged between 18-65 who applied to the AFSÜ PTR Polyclinic and had complaints of neck and back pain for at least 3 months and were diagnosed with myofascial pain syndrome based on anamnesis and physical examination.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — The patients' demographic information, weight and height measurements, occupational activities and desk work time, daily screen usage time, pain intensity (with VAS), cervical joint range of motion examination, pain threshold (with pressure algometer), functional status (with Neck Pain Disability Scale), sleep quality (with Pittsburgh Sleep Quality Scale), anxiety and depression symptoms (with Beck Depression Inventory), cognitive aspects of pain (with Pain Catastrophizing Scale) will be evaluated. The patients' chronotype preferences will be evaluated with Morningness Eveningness Questionnaire.

SUMMARY:
The aim of this study is to examine chronotype preferences in myofascial pain syndrome and to investigate its relationship with pain severity, disability and quality of life.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is defined as sensory, motor, and autonomic symptoms caused by myofascial trigger points. Trigger points are defined as tender points in discrete taut bands of stiffened muscle that cause local and referred pain, among other symptoms. The mechanical and psychological stress of the muscle can activate trigger points and cause pain over a wide area. MyofascialPainSyndrome (MPS) is considered one of the most common chronic musculoskeletal pains. Various studies have shown that it is often associated with depression and anxiety. It is important to focus on modifiable biopsychosocial factors, while paying attention to aspects that cannot be changed, such as attitudes, neuroticism, and trait anxiety, which are known to be somewhat stable over time. Knowing these factors is necessary to improve patients' quality of life and regain their functions.

Pain in patients with MAS can cause sleep disorders such as non-restorative sleep or difficulty initiating or maintaining sleep. It is estimated that 70-80% of patients with MAS experience sleep disorders. Patients with insomnia, especially those living in urban affluent areas, are at risk of developing MAS later in life. Morning-evening preference is an inter-individual difference, also known as diurnal or circadian preference.

The circadian rhythm is controlled by the endogenous circadian clock, which has a genetic basis and is affected by exogenous factors. Due to these individual differences, individuals' energy levels during the day vary so much that people prefer to be active at different times of the day. Morning Type individuals prefer to be active early in the day, while evening type individuals prefer to be active later in the day. Individuals who are between these types and morning or evening preference are called intermediate types. Morning preference is affected by biological factors (e.g., body temperature, cortisol, melatonin), technological and social factors (e.g., electronic media, lighting, TV screens, daily life activities), and environmental factors (e.g., climate, latitude, longitude). In addition, morning preference is related to personality, health, eating habits and psychological well-being. Morning people are more conscientious and more prone to healthy behaviors. On the other hand, evening preference can lead to behavioral problems (e.g., depression, loneliness), personality disorders (substance abuse, eating disorders, internet addiction, daytime sleepiness) and poor academic performance. A study in which 1548 people with fibromyalgia (FMS) were assessed with an online survey that included questions about sleep quality, well-being, pain, chronotype and FMS showed that late chronotypes were more affected by fibromyalgia.

Another study investigating the relationships between chronotypes and musculoskeletal pain showed that evening and intermediate chronotypes were associated with musculoskeletal pain, but mental distress, insomnia, and comorbidities also played a role in these relationships. The aim of this study is to examine chronotype preferences in myofascial pain syndrome and to investigate its relationship with pain severity, disability and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* neck-back pain for at least 3 months
* diagnosis of myofascial pain syndrome by anamnesis and physical examination

Exclusion Criteria:

* Cervical Radiculopathy/Myelopathy
* Recent injection or physical therapy within the last 3 months
* Neck and shoulder surgery
* Neurological and inflammatory diseases
* Pregnancy
* Malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 who applied to Afyonkarahisar Health Sciences University (AFSU) Physical Medicine and Rehabilitation Polyclinic and who have had neck and back pain complaints for at least 3 months were diagnosed with myofascial pain syndrome through anamnesis and physical examination.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
VAS | "Baseline"
  The Visual Pain Scale (VAS), which is easy to understand, apply and interpret, and provides valid and reliable data in a short time, is the most commonly used method in clinics. With a 100 mm visual linear scale, the patient is told that there is no pain at 0, and that the most severe pain they have ever felt at 100, and the patient is asked to put a mark on the point corresponding to their pain.
Pressure Algometry Measurements: (kg/cm2) | "Baseline"
  Algometry measurements will be measured with the Baseline Push Pull Force Gauge ® (Fabrication Enterprises, Inc. PO Box 1500, White Plains, New York 10602, USA) algometry device from the painful trigger point area with the patient in a sitting position.
  Pressure will be applied slowly until the participant first feels pain and responds by saying "stop" and three measurements will be taken with a 30-second interval after each measurement and the average of the three measurements will be recorded as the final value.
Cervical joint range of motion | "Baseline"
  Active passive ROM (flexion, extension, right-left) flexion and rotation) of the cervical joint will be measured.
Morningness Eveningness Questionnaire | "Baseline"
  One of the most widely used tools to assess sleep chronotype preferences. This 19-item screening questionnaire has a rating range of 16 to 86.
  The scoring results are classified as follows: evening types with scores between 16 and 41, morning types with scores between 59 and 86, and no types with scores between 42 and 58.
  The Turkish version has been shown to have good validity and reliability

SECONDARY OUTCOMES:
Neck Pain Disability Scale | "Baseline"
  The questionnaire consists of 20 items and measurements. It includes questions about neck movements, pain intensity, the effect of neck pain on mood, and daily living activities. Each section is scored on a 0-5 rating scale and the total score ranges from 0-100. The Turkish version of this scale was found to be valid and reliable.
Pittsburg Sleep Quality Index (PSQI) | "Baseline"
  PSQI consists of 24 questions in total. 19 of these questions are self-assessment questions. The remaining 5 questions are questions answered by the individual's roommate or spouse, if any. Question 19 on the scale asks whether the participant has a roommate or spouse. The answer to this question is not included in the score calculation. The first 18 questions answered by the participant are used in calculating the total PSQI score and component scores.
  The 18 questions answered by the participant provide information about 7 components: sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), use of sleeping pills (component 6) and daytime sleep dysfunction (component 7). Each component is evaluated on a scale of 0-3 points. The sum of these 7 component scores gives the total PSQI score. The total PSQI score varies between 0-21. The sleep qual
Beck Depression Anxiety Inventory | "Baseline"
  The Beck Depression Inventory is a self-assessment scale consisting of 21 items. Each item is scored between 0 and 3, the highest score that can be obtained from the scale is 63, and the lowest score is 0. A high score from the scale indicates that the severity or level of depression is high.
The Pain Catastrophizing Scale | "Baseline"
  The Pain Catastrophizing Scale is a 13-item self-report inventory using a 5-point Likert scale (0-4) developed by Sullivan et al. to measure the extent to which people catastrophize in response to pain. The original scale consists of three subfactors called helplessness, magnification, and rumination.
SF-12 | "Baseline"
  SF-12 is an easy-to-apply questionnaire with proven reliability and validity, obtained by shortening and simplifying SF-36. It is used to assess the two main components of general health status, physical and mental health. Consisting of twelve questions, SF-12 has mental and physical component scores. High scores indicate good health status.

IPD SHARING:
Plan to Share IPD: No